CLINICAL TRIAL: NCT00722761
Title: A Single-Center, Randomized Double-Blind, Parallel-Group Study to Examine the Safety and Efficacy Of YAZ Compared With Placebo In The Treatment Of Moderate Truncal Acne Vulgaris
Brief Title: Safety and Efficacy Of Drospirenone and Ethinyl Estradiol vs Placebo in the Treatment of Truncal Acne
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Alexandra Kimball, Director, Clinical Unit for Research Trials in Skin, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2008-P-000754
Record Dates: First submitted 2008-07-24; First posted 2008-07-28 (Estimated); Results first posted 2013-03-05 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-01

CONDITIONS: Acne Vulgaris
Keywords: YAZ; oral contraceptive; Acne vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — drospirenone; Ethinyl Estradiol; drospirenone and ethinyl estradiol combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drosperinone and Ethinyl estradiol (Active Comparator): Drospirenone and Ethinyl estradiol (3mg/0.02mg)(YAZ)tablet once a day
  Interventions: Drug: drospirenone and ethinyl estradiol
- Placebo tablet (Placebo Comparator): Placebo tablet once a day
  Interventions: Drug: Placebo tablet

INTERVENTIONS:
Drug: drospirenone and ethinyl estradiol — Drosperinone (3mg) and ethinyl estradiol (0.02mg) tablet given once daily for 24 weeks
  Other Names: YAZ
  Arms: Drosperinone and Ethinyl estradiol
Drug: Placebo tablet — Placebo tablet (no active drug) given once daily for 24 weeks
  Other Names: Placebo
  Arms: Placebo tablet

SUMMARY:
The purpose of this study is to find out if taking a birth control pill, YAZ, is safe and effective for treating acne on the trunk (the main part of the body that does not include the arms, legs, and head).

Acne vulgaris is a very common skin disorder. It is caused when oil-producing skin glands (sebaceous glands) become plugged. The plug can cause blackheads, whiteheads, pimples, and cysts on the face, neck, upper chest, and upper back.

YAZ is a combination birth control pill. A "combination" pill means that it is made up of more than one major ingredient. Nearly all birth control pills are made up of a combination of estrogen and progestin hormones. Estrogens are steroid hormones produced by the ovaries responsible for the typical female features. Progestins are steroid hormones produced by the ovary and placenta responsible for making the uterus fit for pregnancy. YAZ also contains an estrogen called ethinyl estradiol, and a progestin called drospirenone. People who develop acne have sebaceous glands that are over-stimulated (that is, the sebaceous glands have increased activity) by male sex hormones (androgens). The progestin in YAZ blocks the male sex hormones (androgens) that cause acne.

The study drug being used in this study is called YAZ. It has been approved by the U.S. Food and Drug Administration (FDA) to treat moderate acne in women who want an oral contraceptive for birth control.

In this study, YAZ will be compared to a placebo for safety and effectiveness. A placebo looks like the study drug but contains no active drug (like a sugar pill). We use placebos in research studies to learn if the effects seen in research subjects are truly from the study drug or from other reasons.

DETAILED DESCRIPTION:
Acne is a common skin disease that affects 85-100% of the population. Although it often appears during puberty, it may persist during the third decade of life and even later. It is characterized by a variety of lesions consisting of non-inflammatory lesions known as comedones, and inflammatory lesions such as papules, pustules, nodules and cysts. It commonly occurs on the face, chest, and back. Although not as noticeable as facial acne, truncal acne may also affect a person's self esteem and body image and reduce one's participation in sports because of the need to undress in a shared locker room. Most acne studies focus on facial acne and ignore treatment outcomes in the chest and back.

The pathogenesis of acne is multifactorial, developing in the sebaceous gland. These factors include intrafollicular hypercornification, which induces follicular obstruction resulting in comedone formation, excess sebum production, Propionibacterium acnes activity and inflammation.

Hormone therapies, such as oral contraceptives and antiandrogens (e.g. spironolactone) counteract the effects of androgens on the sebaceous glands. It has been over ten years since estrogen-containing oral contraceptives (OCs) first obtained FDA approval for use in acne. Since then, several randomized controlled trials have corroborated their efficacy and safety for this growing indication in women of child bearing age. Studies have shown hormonal therapies to be effective in treating moderate acne vulgaris in women with no known contraindication to OC therapy.

YAZ is an oral contraceptive that is FDA approved for acne vulgaris. Unlike other progestins, drospirenone has unique antimineralocorticoid (mild diuretic effect) and antiandrogenic properties. The antiandrogenic property of drospirenone means that it blocks the male sex hormones that can cause acne. In two multicenter, double blind, randomized, placebo-controlled studies, 889 subjects, ages 14 to 45 years, with moderate acne received YAZ or placebo for six 28 day cycles. The primary efficacy endpoints were the percent change in inflammatory lesions, non-inflammatory lesions, total lesions, and the percentage of subjects with a "clear" or "almost clear" rating on the Investigator's Static Global Assessment (ISGA) scale on day 15 of cycle 6.

Subjects will be assigned to a treatment group upon randomization. Bayer HealthCare Pharmaceuticals personnel, investigators, subjects and study nurse/coordinators will be blinded to the study product treatment assignment. The study duration will be 24 weeks with visits at screening, baseline (week 0), week 6, week 12, week 18, and week 24. Lesion counts (total, inflammatory, non-inflammatory) and an ISGA, and photography will be performed on every visit. A physical examination will be done at baseline and Week 24. Safety will be assessed from reported adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

* Female Subjects 18-45 years of age who have achieved spontaneous menarche.
* A clinical diagnosis of truncal acne vulgaris and the desire for an oral contraceptive for birth control.
* A minimum of 10 but not more than 50 inflammatory lesions on the back and chest combined.
* Maximum of 5 nodules.
* Willing and able to understand and sign informed consent.
* Able to complete study and comply with study procedures.

Exclusion Criteria:

* Use of topical acne medications such as tretinoin, benzoyl peroxide or topical antibiotics within 2 weeks
* Use of oral antibiotics within 30 days.
* Use of systemic corticosteroids within 4 weeks.
* Use of oral contraceptives within 12 weeks.
* Use of isotretinoin in past six months.
* Use of phototherapy devices for acne such as ClearLight or Zenozapper within 1 week.
* Use of tanning booths or lamps within 1 week prior to baseline.
* BMI >30
* History of renal insufficiency
* History of hepatic dysfunction
* History of adrenal Insufficiency
* History of vascular or metabolic disease including existing or previous arterial thromboembolic diseases (myocardial infarction, stroke), existing or previous venous thromboembolic diseases (deep vein thrombosis, pulmonary embolism), and any condition which could increase the risk to suffer any of the above mentioned disorders
* History of hypertension
* Diabetes mellitus with vascular involvement
* Migraine headaches with focal neurological symptoms
* Recent major surgery with prolonged immobilization
* Known or suspected carcinoma of the breast
* Carcinoma of the endometrium or other known or suspected estrogen-dependent neoplasia
* Undiagnosed abnormal genital bleeding
* Cholestatic jaundice of pregnancy or jaundice with prior pill use
* Liver tumor (benign or malignant) or active liver disease
* Smoking > ½ pack of cigarettes/week
* Regular intake of medications that may increase potassium levels such as NSAIDS, potassium sparing diuretics, potassium supplementation, ACE inhibitors, Angiotensin-II receptor antagonists, heparin and aldosterone antagonists.
* Hypersensitivity to any component of the study drug
* Clinically significant abnormal findings or conditions (other than acne), which might, in the opinion of the Principal Investigator, interfere with study evaluations or pose a risk to subject safety during the study.
* Subjects who are known to be pregnant or planning a pregnancy.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra B. Kimball, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Clinical Unit for Research Trials in Skin, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Females, age 18 to 45 years, who achieved spontaneous menarche and had a diagnosis of truncal acne of 10 to 50 inflammatory lesions on the back and chest combined with not more than 5 nodules
Groups:
- Drosperinone and Ethinyl Estradiol: Drospirenone (3mg) and Ethinyl estradiol (0.02mg) (YAZ)tablet once a day
Period: Overall Study
Arm/Group | Drosperinone and Ethinyl Estradiol | Placebo Tablet
Started | 16 | 14
COMPLETED AT LEAST 1 FOLLOW-UP VISIT | 15 | 10
Completed | 10 | 8
Not Completed | 6 | 6
Not completed — Lost to Follow-up | 1 | 4
Not completed — Withdrawal by Subject | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Drosperinone and Ethinyl Estradiol | Placebo Tablet | Total
Number analyzed (Participants) | 16 | 14 | 30
Age Continuous [Mean (Standard Deviation); unit: years] | 23 (5.1) | 24 (3.7) | 24 (4.5)
Sex/Gender, Customized [Number; unit: participants]
  Female | 16 | 14 | 30
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 1 | 0 | 1
  Asian | 2 | 2 | 4
  African American | 2 | 1 | 3
  Caucasian | 11 | 11 | 22
BMI [Mean (Standard Deviation); unit: kg/m2] | 23.2 (2.2) | 23.6 (2.6) | 23.4 (2.9)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Truncal Lesion Counts
Description: Acne lesion count (noninflammatory, inflammatory and total lesions) difference between week 0 (baseline) and week 24 is divided by the acne lesion count at week 0 and multiplied by 100. A positive change indicates a decrease in truncal acne lesions.
Time Frame: 0-24 weeks
Population: Intention to treat analysis. Only participants with at least one follow up were included in the analysis. Last observation carried forward was used to fill up missing data.
Measure: Mean (Standard Deviation); unit: percentage change of lesions
Arm/Group | Drosperinone and Ethinyl Estradiol | Placebo Tablet
Number analyzed (Participants) | 15 | 10
percentage change of lesions
  Noninflammatory lesions | 52.1 (43.3) | -9.2 (77.6)
  Inflammatory lesions | 53.2 (40.9) | 18.2 (40.1)
  Total acne lesions | 51.8 (31.9) | 17 (47.1)

2. Secondary Outcome: Percentage of Subjects Rated Clear or Almost Clear on the IGA and SGA at Week 24/ Early Termination
Description: Percentage of subjects rated Clear (score 0) or Almost Clear (score 1) on the Investigator's Global Assessment (IGA) of truncal acne at Week 24 as well as Subject's Assessment of Acne at Week 24/Early Termination were taken. It was computed by: number of successes (those scored 0 or 1)divided by the number of participants multiplied by 100.
Time Frame: 24 weeks
Population: Intention to treat analysis. Participants with at least one follow up visit were included in the analysis. Last observation carried forward was used to fill up missing values/
Measure: Number; unit: percentage of participants
Arm/Group | Drosperinone and Ethinyl Estradiol | Placebo Tablet
Number analyzed (Participants) | 15 | 10
percentage of participants
  Investigator Global Assessment IGA | 53.3 | 20
  Subject Assessment SGA | 60 | 80

ADVERSE EVENTS:
Arm/Group | Drosperinone and Ethinyl Estradiol | Placebo Tablet
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14
Other Adverse Events (participants affected / at risk) | 2/16 | 0/14
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drosperinone and Ethinyl Estradiol (N=16) | Placebo Tablet (N=14)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Loss of appetite (Nervous system disorders) | 1 (1) | 0 (0)
moodiness (Nervous system disorders) | 1 (1) | 0 (0)
break through bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination leading to small number of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No